CLINICAL TRIAL: NCT01586949
Title: A Randomized Controlled Trial of the Effectiveness of the Web-based Well-being Intervention Daily Challenge
Brief Title: Effectiveness of a Well-being Web-based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MeYou Health, LLC (Industry)
Collaborators: Healthways, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DC-EFF-2012
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Focus of Study: Healthy Individuals
Keywords: well-being; web-based intervention; social networks

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Intervention: Daily Challenge
  Interventions: Behavioral: Daily Challenge
- Control (No Intervention): Weekly Well-being, an email-based health information delivery service.

INTERVENTIONS:
Behavioral: Daily Challenge — Web-based behavioral intervention aiming to improve individuals' well-being.
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine whether the intervention Daily Challenge (MeYou Health, LLC), a behavioral intervention delivered online, is effective in improving individuals' well-being.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older, 19 years of age or older if participant resides in Alabama or Nebraska)
* Provided informed consent to participate in the study

Exclusion Criteria:

* Does not live in the United States of America
* Has a Facebook friend enrolled in the study
* Fails to complete the informed consent and registration process in the allotted time (45 minutes)
* Gender (recruitment will be titrated to ensure a minimum of 30% male ratio)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1503 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Well-being score, as determined by the Healthways Well-Being Assessment | Baseline, 30 days, 90 days
  Change in well-being score

SECONDARY OUTCOMES:
Interpersonal support score, as evaluated with the Interpersonal Support Evaluation List (ISEL) | Baseline, 30 days, 90 days
  Change in interpersonal support score.

CONTACTS AND LOCATIONS:
Overall Officials: Josee Poirier, PhD, Principal Investigator — MeYou Health, LLC; Nathan K Cobb, MD, Study Chair — MeYou Health, LLC
Locations (1):
- MeYou Health office, Boston, Massachusetts, United States

REFERENCES:
- [Background] Harrison PL, Pope JE, Coberley CR, Rula EY. Evaluation of the relationship between individual well-being and future health care utilization and cost. Popul Health Manag. 2012 Dec;15(6):325-30. doi: 10.1089/pop.2011.0089. Epub 2012 Feb 22. PMID 22356589
- [Background] Prochaska JO, Evers KE, Castle PH, Johnson JL, Prochaska JM, Rula EY, Coberley C, Pope JE. Enhancing multiple domains of well-being by decreasing multiple health risk behaviors: a randomized clinical trial. Popul Health Manag. 2012 Oct;15(5):276-86. doi: 10.1089/pop.2011.0060. Epub 2012 Feb 21. PMID 22352379
- [Background] Heesch KC, Masse LC, Dunn AL, Frankowski RF, Mullen PD. Does adherence to a lifestyle physical activity intervention predict changes in physical activity? J Behav Med. 2003 Aug;26(4):333-48. doi: 10.1023/a:1024205011001. PMID 12921007
- [Background] Strecher VJ, McClure J, Alexander G, Chakraborty B, Nair V, Konkel J, Greene S, Couper M, Carlier C, Wiese C, Little R, Pomerleau C, Pomerleau O. The role of engagement in a tailored web-based smoking cessation program: randomized controlled trial. J Med Internet Res. 2008 Nov 4;10(5):e36. doi: 10.2196/jmir.1002. PMID 18984557
- [Background] Hill JO, Wyatt HR, Reed GW, Peters JC. Obesity and the environment: where do we go from here? Science. 2003 Feb 7;299(5608):853-5. doi: 10.1126/science.1079857. PMID 12574618
- [Background] Hill JO. Can a small-changes approach help address the obesity epidemic? A report of the Joint Task Force of the American Society for Nutrition, Institute of Food Technologists, and International Food Information Council. Am J Clin Nutr. 2009 Feb;89(2):477-84. doi: 10.3945/ajcn.2008.26566. Epub 2008 Dec 16. PMID 19088151
- [Background] Eysenbach G. The law of attrition. J Med Internet Res. 2005 Mar 31;7(1):e11. doi: 10.2196/jmir.7.1.e11. PMID 15829473
- [Background] Christakis NA. Social networks and collateral health effects. BMJ. 2004 Jul 24;329(7459):184-5. doi: 10.1136/bmj.329.7459.184. No abstract available. PMID 15271805
- [Background] Christakis NA, Fowler JH. The spread of obesity in a large social network over 32 years. N Engl J Med. 2007 Jul 26;357(4):370-9. doi: 10.1056/NEJMsa066082. Epub 2007 Jul 25. PMID 17652652
- [Background] Christakis NA. Health care in a web. BMJ. 2008 Jun 28;336(7659):1468. doi: 10.1136/bmj.a452. PMID 18583678
- [Background] Pew Research Center. Social networking sites and our lives (Report). 2011. http:/pewinternet.org/Reports/2011/Technology-and-social-networks.aspx
- [Background] Helliwell JF, Putnam RD. The social context of well-being. Philos Trans R Soc Lond B Biol Sci. 2004 Sep 29;359(1449):1435-46. doi: 10.1098/rstb.2004.1522. PMID 15347534
- [Background] Stata analysis software. Stata Corporation, College Station, TX.
- [Background] Tabachnick, B.G. and Fidell, L.S. Using multivariate statistics, 4th Edition, Allyn & Bacon, Needham, MA. 2001.
- [Background] Fleiss, J.L. Design and Analysis of Clinical Experiments.1999. Wiley, New York, NY.
- [Background] MacKinnon DP, Fairchild AJ, Fritz MS. Mediation analysis. Annu Rev Psychol. 2007;58:593-614. doi: 10.1146/annurev.psych.58.110405.085542. PMID 16968208
- [Background] Beasley, T.M. Seemingly unrelated regression (SUR) models as a solution to path analytic models with correlated errors. Multiple Linear Regression Viewpoints. 34(1): 1-7, 2008.
- [Background] Zellner, A. An efficient method of estimating seemingly unrelated regressions and tests for aggregation bias. J Am Stat Assoc, 57(348-68), 1962.
- [Background] Lin DY, Fleming TR, De Gruttola V. Estimating the proportion of treatment effect explained by a surrogate marker. Stat Med. 1997 Jul 15;16(13):1515-27. doi: 10.1002/(sici)1097-0258(19970715)16:133.0.co;2-1. PMID 9249922
- [Background] Vittinghoff E, Sen S, McCulloch CE. Sample size calculations for evaluating mediation. Stat Med. 2009 Feb 15;28(4):541-57. doi: 10.1002/sim.3491. PMID 19065627
- [Background] Gleason, T.C. and Staelin, R. A proposal for handling missing data. Psychometrika, 40(2): 229-252, 1975.
- [Background] Little, R.J. and Rubin, D.B. Statistical analysis with missing data, 2nd Edition, Wiley, New York, NY. 2002.
- [Background] Schafer, J. L. Analysis of Incomplete Multivariate Data. New York, NY: Chapman & Hall, CRC. 2002.
- [Derived] Cobb NK, Poirier J. Effectiveness of a multimodal online well-being intervention: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):41-8. doi: 10.1016/j.amepre.2013.08.018. PMID 24355670